CLINICAL TRIAL: NCT04364633
Title: Study of the Impact of a Intra-tracheal Intubation With Curarization or Without Curarization (With Remifentanil) on the Self-perception of the Voice.
Brief Title: Impact of a Intra-tracheal Intubation With Curarization or Without Curarization
Acronym: VHIntubation
Status: Terminated | Type: Observational
Why Stopped: Premature termination of the study because it was dependent on the Remicrush study which ended more quickly, not allowing the inclusion of the expected number of patients.
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC20_0058
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2021-09

CONDITIONS: Intubation Complication
Keywords: Intra-tracheal intubation; Voice Handicap; Remifentanil; Curarization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Remifentanil group: bolus intravenous injection of 3 to 4µg/kg of remifentanil after hypnotic administration for a crush anesthetic induction
  Interventions: Other: Voice Handicap Questionnaire (VHI)
- Neuromuscular blockade group: Bolus intravenous injection of 1mg/kg of Succinylcholine or Rocuronium after hypnotic administration for a crush anesthetic induction
  Interventions: Other: Voice Handicap Questionnaire (VHI)

INTERVENTIONS:
Other: Voice Handicap Questionnaire (VHI) — Voice Handicap Index (VHI) self-questionnaire

SUMMARY:
VHIntubation is a French monocentric and observational study that will assess the impact of two intra-tracheal intubation preparation procedures (curarization versus remifentanil) on the voice, using the Voice Handicap Index (VHI) self-questionnaire.

DETAILED DESCRIPTION:
Some surgeries are known to expose patients to voice disorders (thyroidectomy, parathyroidectomy, carotid surgery…). However, voice disorders can be due, among other things, to a laryngeal nerves alteration and intubation trauma. Our team has published 2 prospective studies on the frequency of voice troubles after thyroidectomy (Borel et al. Surgery 2018 and 2019).

To limit post tracheal intubation voice troubles , it is generally recommended to practice intra-tracheal intubation with a curarization (Lundstrøm et al. Br J Anaesth 2018). However, for few years, the very vast majority of thyroid surgery is practiced with a neuromonitoring of laryngeal nerves (NIM). NIM ensures prosper functioning of the vocal cords intra- and post-operatively with an excellent negative predictive value (>98%, Mirallié et al. Surgery 2018). However, the use of NIM requires an absence of curarization. Some centres, including ours, have abandoned systematic curarization before intubation for thyroidectomy; other centres continue to practice curarization with, sometimes, the need to antagonize curarization for an effective NIM utilization.

The aim of this study is to assess the impact of intubation preparation procedures (curarization versus remifentanil) on the voice using Voice Handicap Index (VHI) questionnaire.

The Nantes University Hospital is the sponsor of " REMICRUSH ", study on " Assessment of Remifentanil for Rapid Sequence Induction and Intubation in Full Stomach Patient Compared to Muscle Relaxant. A Non-inferiority Simple Blind Randomized Controlled Trial ", the coordinator of which is Dr Nicolas Grillot.

This study began in October 2019 and authorisations are obtained. We aim to propose our study " VHIntubation " to patients participating in REMICRUSH in order to benefit from REMIFENTANIL versus CURARE randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in " REMICRUSH " study
* patient's non-opposition to participation in research

Inclusions criteria in REMICRUSH are :

* male or female aged from 18 to 80 years old
* surgery requiring general anaesthesia with tracheal with oro-tracheal intubation
* Rapid sequence intubation indication
* aspiration risk defined as : fasting < 6h00, digestive occlusion, functional ileus, vomiting < 12h00, orthopaedic trauma < 12h00, severe gastric reflux, gastroparesis and/or dysautonomia and or gastro-oesophagus surgery
* signed informed consent sheet ; or emergency procedure if impossible

Exclusion Criteria:

* Patients non-included in " REMICRUSH " study
* Patients with cervical surgery
* Patient declines to participate in research

Exclusion criteria in REMICRUSH are :

* planned impossible intubation
* suspected/known allergy to neuromuscular blockade or remifentanil
* neuromuscular disease forbidding neuromuscular blockade use
* Prolonged neuromuscular block former episode
* Malignant hyperthermia former episode
* Pre-operative respiratory failure (spO2< 95%)
* Pre-operative hemodynamic failure (use of vasopressor) cardiac arrest
* A woman of childbearing age who has an active pregnancy and/or clinical signs suggestive of an active pregnancy and/or does not have a contraceptive or contraceptive method and has had unprotected sex within 15 days of the last menstrual period.
* Patients under justice protection
* Use of etomidate for anesthetic induction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Nantes University Hospital is the sponsor of " REMICRUSH ", study on " Assessment of Remifentanil for Rapid Sequence Induction and Intubation in Full Stomach Patient Compared to Muscle Relaxant. A Non-inferiority Simple Blind Randomized Controlled Trial ", We aim to propose our study " VHIntubation " to patients participating in REMICRUSH in order to benefit from REMIFENTANIL versus CURARE randomization.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Voice Handicap at 1 month post-intubation | 1 month post-intubation
  Evaluate the impact of the procedures to prepare at intra-tracheal intubation (curarization versus remifentanil) on the voice, using Voice Handicap Index (VHI) self-questionnaire at 1 month post-intubation.
  Primary endpoint is the evolution of the score at VHI questionnaire (Voice Handicap Index) at 1 month post-intubation, the reference is the pre-intubation score. An augmentation of 18 points score is considered as significant (Borel et al. Surgery 2018).

SECONDARY OUTCOMES:
Voice Handicap at 6 month post-intubation | 6 month post-intubation
  Evaluate the impact of the procedures to prepare at intra-tracheal intubation (curarization versus remifentanil) on the voice, using Voice Handicap Index (VHI) self-questionnaire at 6 month post-intubation.
  Primary endpoint is the evolution of the score at VHI questionnaire (Voice Handicap Index) at 6 month post-intubation, the reference is the pre-intubation score. An augmentation of 18 points score is considered as significant (Borel et al. Surgery 2018).

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France